CLINICAL TRIAL: NCT00587665
Title: A Prospective Study of Low Dose Ketamine as an Adjunct to Fentanyl in Pediatric Patients Following Outpatient Tonsillectomy and Adenoidectomy
Brief Title: Low Dose Ketamine as an Adjunct to Fentanyl in Outpatient Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Gregory J. Schears, MD, Mayo Clinic, Rochester, MN
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1896-05
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2007-12

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Low dose ketamine given
  Interventions: Drug: ketamine
- 2 (Placebo Comparator): Saline given as control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ketamine — Single IV dose of 0.1 mg/kg of ketamine
  Arms: 1
Drug: Placebo — Saline given of equal volume to drug
  Arms: 2

SUMMARY:
Comparing patients receiving subanesthetic doses of Ketamine vs placebo to see if it can reduce narcotic needs for patients receiving a tonsillectomy and adenoidectomy

ELIGIBILITY:
Inclusion Criteria:between 3 and 12 years of age

* ASA 1 or 2

Exclusion Criteria:

* did not consent

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
amount of post op narcotic use | 5 days

SECONDARY OUTCOMES:
degree of nausea and vomiting | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Schears, md, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States